CLINICAL TRIAL: NCT06317454
Title: Genetic and Environmental Determinants of Metabolic Control in Children and Young Adults With Type 1 Diabetes Mellitus
Brief Title: Determinants of Metabolic Control in Children With Type 1 Diabetes Mellitus
Status: Recruiting | Type: Observational
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: GR-2019-12369573
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 diabetes; Metabolic control
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects with T1DM
  Interventions: Diagnostic Test: Blood and saliva analysis
- Control subjects
  Interventions: Diagnostic Test: Blood and saliva analysis

INTERVENTIONS:
Diagnostic Test: Blood and saliva analysis — Phenotyping and genotyping characterization using blood and saliva

SUMMARY:
A good metabolic control of type 1 diabetes mellitus (T1DM) is crucial to avoid long-term complications associated with the disease. Although recent evidences suggest that a good metabolic control of T1DM is partly independent of management intensity and could be anticipated since onset, factors that influence glycated haemoglobin (HbA1c) patterns remain poorly understood and are likely to be genetic.

While significant progress has been made in understanding of the genetic contribution to T1DM onset, very few studies have evaluated the role of genetic factors on T1DM metabolic control.

This study aims to create a comprehensive database of genetic and phenotypic data in a cohort of children and young adults with T1DM and to evaluate genetic and environmental factors that might predict trajectories in glycemic control

ELIGIBILITY:
Inclusion Criteria

Cases:

* age between 6 and 21 years;
* patients suffering from type 1 diabetes

Controls:

* age between 6 and 21 years;
* patients for whom a venous sampling is planned

Exclusion criteria

Cases:

* patients for whom it is not possible to collect information on the clinical history, starting from the onset of diabetes
* patients with other types of diabetes mellitus (type 2, monogenic diabetes, diabetes related to cystic fibrosis...)
* patients incapable of expressing valid informed consent or whose parents are incapable of expressing valid informed consent.

Controls:

* subjects with type 1 and 2 diabetes
* obese subjects and those with a family history of diabetes and obesity or other metabolic disorders
* subjects with HbA1c >6%
* patients incapable of expressing valid informed consent or whose parents are incapable of expressing valid informed consent.

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients between 6 and 21 years with or without type 1 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of environmental factors affecting T1DM metabolic control | Through study completion, an average of 18 months
Identification of genetic factors affecting T1DM metabolic control | Through study completion, an average of 18 months
  Identify genetic factors responsible of differences in T1DM metabolic control and thus uncover genes of potential biological therapeutic importance

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Maternal and Child Health - IRCCS "Burlo Garofolo", Trieste, Italy